CLINICAL TRIAL: NCT02551328
Title: A Single-center Observational Study Investigating the Effect of Volatile Conditioning (VC) With Sevoflurane on Myocardial Biomarkers and Platelets Function in Patients Having Minimally Invasive Mitral Valve Surgery (MIMV)
Brief Title: Preconditioning With Sevoflurane and Propofol in Patients Undergoing Minimally Invasive Mitral Valve Surgery
Acronym: MINI-SEVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Responsible Party: Principal Investigator, MOSCARELLI MARCO, MD, PhD, Fondazione Toscana Gabriele Monasterio
Other Study IDs: 452/2014
Record Dates: First submitted 2015-09-01; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sevofluorane: Patients preconditioned with Sevo
  Interventions: Drug: sevofluorane
- Propofol: Patients with no preconditioning

INTERVENTIONS:
Drug: sevofluorane — Continuous infusion of sevofluorane
  Other Names: SEVO
  Groups: Sevofluorane

SUMMARY:
The main aim of this study is to compare markers of cardiac injury (Troponin I), inflammatory response and platelets function during minimally invasive mitral valve repair or replacement (MIMV) via right mini-thoracotomy in two standard anaesthetic regimes (sevo \propofol)

DETAILED DESCRIPTION:
The main aim of this study is to compare markers of cardiac injury (Troponin I), inflammatory response and platelets function during minimally invasive mitral valve repair or replacement (MIMV) via right mini-thoracotomy in two standard anaesthetic regimes:

* Volatile conditioning (sevoflurane) used during induction (preconditioning) and during the operation as maintenance (perconditioning) and no propofol.
* Propofol induction and maintenance (TIVA) and no volatile anaesthetics.

Outlet/residual blood samples coming from routine check will be collected at different time points.

Study will be powered on Troponin I (primary statistical outcome). Original secondary outcome will be considered: platelets activation, left ventricle function, clinical figures (length of stay, inotrops requirements, ventilation times and other relevant).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Patients undergoing elective (or urgent) first-time minimal invasive mitral valve surgery.

Exclusion Criteria:

1. Cardiogenic shock or cardiac arrest, emergent CABG
2. Renal failure (with a GFR < 30 ml/min/1.73m2),
3. Glibenclamide or nicorandil (as these medications may interfere with VC)
4. Pregnancy
5. Known intolerance/allergy to sevoflurane or propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age>=18 Pt undergoing elective (or urgent) first-time minimal invasive mitral valve surgery Pt will have to sign informed consent
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Myocardial Injury assessed by changes in Troponin values | properatively-6, 12, 24, 48 and 72 hours after the end of ischaemic cardioplegic arrest
  According to the routine post operative blood testing frame-time troponin sample will collected in the preoperative and postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Del Sarto, MD, Principal Investigator — Fondazione Toscana Gabriele Monasterio
Locations (1):
- Ospedale del cuore, Pasquinucci Hospital, Fondazione Monasterio, Massa, Italy, Italy